CLINICAL TRIAL: NCT02695966
Title: A Feasibility Study Assessing the Ability of an Ex-vivo Assay to Measure AMD3100's Ability to Overcome Tumour Immune-privilege and Bring T-lymphocytes Into Contact With Neoplastic Targets.
Brief Title: EVIS - Ex-vivo Assessment of T-lymphocyte Homing in Primary Pancreatic Cancer
Acronym: EVIS
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Cancer Research UK Cambridge Institute (Other); University of Cambridge (Other)
Responsible Party: Principal Investigator, CCTU- Cancer Theme, Clinical Trial Coordinator, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: EVIS
Record Dates: First submitted 2016-02-23; First posted 2016-03-02 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour tissue sample Blood sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Whipples Surgery — Whipples Surgery

SUMMARY:
This is a single-centre, prospective, non-randomised research study. The research team will investigate the feasibility of assessing primary human pancreatic tissue for changes to T lymphocyte function and localisation in the presence and absence of AMD3100.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of cancer-related deaths in Western countries. It is a lethal disease that typically presents late, metastasises early and is resistant to conventional treatments such as radiation and chemotherapy. In 2012 there were 8700 deaths in the UK from pancreatic cancer, making it the fifth most common cause of cancer-related death.

Current therapeutic strategies are aimed at extending survival as well as improving symptoms and quality of life, but although conventional chemotherapeutic agents have achieved modest clinical benefit, the need for novel therapies is great.

This study proposes to extend our pre-clinical studies to develop an ex-vivo assay for the assessment of AMD3100 effectiveness in human samples.

The research team will investigate the feasibility of assessing primary human pancreatic tissue for changes to T lymphocyte function and localisation in the presence and absence of AMD3100 through obtaining a blood sample and fresh pancreatic tissue intra-operatively from pancreatic tumours located in the head of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary pancreatic adenocarcinoma who are undergoing pancreaticoduodenectomy (Whipple's) resection.
* Patients who are over 18 years of age at the time of signing the informed consent form and who are physically and mentally capable of consenting.
* Willing and able to comply with study procedures.

Exclusion Criteria:

• Any condition or abnormalities that in the judgment of the investigator/surgeon/ histopathologist would place the patient at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary pancreatic adenocarcinoma who are undergoing pancreaticoduodenectomy (Whipple's) resection.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Cancer cell distribution | 12 months
  Tumour tissue analysis
T lymphocyte changes | 12 months
  DNA, RNA and protein tumour tissue analysis

SECONDARY OUTCOMES:
T lymphocyte localisation | 12 months
  Tumour tissue analysis using study drug and other agents

CONTACTS AND LOCATIONS:
Overall Officials: James Dr Thaventhiran, Study Chair — University of Cambridge
Locations (1):
- Addenbrooke's Hospital, Cambridge, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No